CLINICAL TRIAL: NCT04791995
Title: REsuscitation and CAPillary rePerfusion - A Cohort Study With Prospective Inclusion
Brief Title: Resuscitation and Capillary Reperfusion
Acronym: ReCapp
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Michael Holzer, Prof. Michael Holzer, Medical University of Vienna
Other Study IDs: 001
Record Dates: First submitted 2021-03-02; First posted 2021-03-10 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Cardiac Arrest; Cardiac Arrest, Out-Of-Hospital; Cardiopulmonary Arrest; Cardiopulmonary Arrest With Successful Resuscitation
Keywords: capillary refill time; skin mottling score; capillary lactate; microperfusion; cardiopulmonary resuscitation
MeSH Terms: conditions — Heart Arrest; Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Persistent microperfusion alterations after return of spontaneous circulation (ROSC) are associated with poor survival. To our knowledge, no human studies evaluating microperfusion during cardiopulmonary resuscitation (CPR) with simple and pre-hospital available tests have been published. Capillary refill time (CRT) and skin-mottling-score (SMS) are parameters for microperfusion and evaluated in septic and cardiogenic shock. In animal studies, microperfusion was impaired during cardiac arrest, although not correlating with systemic blood pressure.

The aim of this study is to investigate the correlation between impaired microcirculation (as measured with CRT and SMS) during resuscitation and ROSC resp. neurological outcome. Our clinical impression in daily routine is, that the appearance of a patient undergoing CPR is often linked to the outcome. We hypothesize, that this is due to changes in microperfusion of the skin.

ELIGIBILITY:
Inclusion Criteria:

* All patients ≥18 years during cardiopulmonary resuscitation
* witnessed cardiac arrest

Exclusion Criteria:

* insufficient manpower (e.g. study team has to provide CPR)
* hypovolemia (exsanguination, anaphylaxis, sepsis as underlying cause)
* presumed or known COVID-19 disease
* hypo-/hyperthermia (<36.0°, >37.5°C)
* Raynaud's disease
* Peripheral arterial disease

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult out-of-hospital cardiac arrest patients
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Capillary refill time (CRT) | baseline (immediately after inclusion to the study)
  Capillary refill time in seconds measured on one finger and one earlobe for ROSC vs. no ROSC

SECONDARY OUTCOMES:
Skin mottling score (SMS) | baseline (immediately after inclusion to the study = minute 0), minute 2, 4, 6, 8, (...) up to return of spontaneous circulation or death, whichever came first
  Skin mottling score (Ait-Oufella, H., Lemoinne, S., Boelle, P.Y. et al. Mottling score predicts survival in septic shock. Intensive Care Med 37, 801-807 (2011). Best: 0 - no mottling to worst: 5 - mottling on the entire leg) for ROSC vs. noROSC
Capillary blood lactate (Lac) | baseline (immediately after inclusion to the study, = minute 0), minute 4, 8, 12, 16, 20
  Capillary lactate in mmol/L from the capillary bed of a finger for ROSC vs noROSC and for correlations with CRT, SMS
Hospital mortality | baseline (immediately after inclusion to the study)
  Correlation of CRT, SMS and Lac with hospital mortality
Correlation of CRT, SMS and Lac and 30 days good neurological outcome | baseline (immediately after inclusion to the study)
  Good neurological outcome at 30 days measured with Cerebral Performance Category (CPC 1-5 (1 best: good cerebral performance, 5 worst: brain dead), modified Rankin scale (mRs 0-6 (0 best: no symptoms, 6 worst: dead) and health utility index 3 (HUI-3, worst: -0,36 - best: 1)
Correlation of CRT, SMS and Lac and hospital discharge good neurological outcome | baseline (immediately after inclusion to the study)
  Good neurological outcome at hospital discharge measured with Cerebral Performance Category (CPC 1-5 (1 best: good cerebral performance, 5 worst: brain dead), modified Rankin scale (mRs 0-6 (0 best: no symptoms, 6 worst: dead) and health utility index 3 (HUI-3, worst: -0,36 - best: 1)
Correlation of CRT/SMS and lactate | baseline (immediately after inclusion to the study)
  Correlation of CRT/SMS and lactate
Correlation of SMS and CRT | baseline (immediately after inclusion to the study)
  Correlation of SMS and CRT
Correlation of time since cardiac arrest and CRT/SMS/lactate | baseline (immediately after inclusion to the study)
  Correlation of time since cardiac arrest and CRT/SMS/lactate
Correlation of catecholamine demand during the first 48 hours after ROSC and CRT/SMS | from ROSC up to 48 hours after ROSC
  Cumulative catecholamine demand during the first 48 hours after ROSC in correlation with CRT/SMS/Lac during resuscitation
Capillary refill time (CRT) | minute 2, 4, 6, 8, (...) up to return of spontaneous circulation or death, whichever came first
  Capillary refill time in seconds measured on one finger and one earlobe for ROSC vs. no ROSC

CONTACTS AND LOCATIONS:
Overall Officials: Michael Holzer, MD, Principal Investigator — Department of Emergency Medicine, Medical University of Vienna
Locations (1):
- Vienna Municipal Emergency Service, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mueller M, Holzer M, Losert H, Grassmann D, Ettl F, Gatterbauer M, Magnet I, Nuernberger A, Kienbacher CL, Gelbenegger G, Girsa M, Herkner H, Krammel M. The association of capillary refill time and return of spontaneous circulation during out-of-hospital cardiac arrest: an observational study. Crit Care. 2025 Jan 21;29(1):37. doi: 10.1186/s13054-025-05255-4. PMID 39838473